CLINICAL TRIAL: NCT00763997
Title: Study of the Effect of Dipyrone, Ibuprofen, Paracetamol and Parecoxib on the Platelet Aggregation
Brief Title: Study of the Effect of Dipyrone, Ibuprofen, Paracetamol and Parecoxib on the Platelet Aggregation in Analgetic Dosages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Matthias Schmauß, MD, scientific associate with the Ruhr Unievrsity Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NRA3480005
Record Dates: First submitted 2008-09-29; First posted 2008-10-01 (Estimated); Last update posted 2008-10-01 (Estimated); Status verified 2008-09

CONDITIONS: Platelet Aggregation
Keywords: dipyrone; platelet aggregation; neuraxial blockage; ibuprofen; platelet aggregation under dipyrone compared to ibuprofen, acetaminophen and parecoxib/valdecoxib; neuraxial blockage in patients receiving ibuprofen is critical in special circumstances, but traditionally not fpr dipyrone
MeSH Terms: interventions — Dipyrone; Ibuprofen; Acetaminophen; parecoxib; valdecoxib; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Dipyrone
  Interventions: Drug: dipyrone; Other: Blood samples
- 2 (Active Comparator): Ibuprofen
  Interventions: Drug: Ibuprofen; Other: Blood samples
- 3 (Active Comparator): Acetaminophen
  Interventions: Drug: Acetaminophen; Other: Blood samples
- 4 (Placebo Comparator): Parecoxib/Valdecoxib
  Interventions: Drug: Parecoxib/Valdecoxib; Other: Blood samples

INTERVENTIONS:
Drug: dipyrone — Dipyrone is given in the operation room with 2,5 g intravenously, followed by an oral regime of 4x1g on the ward
  Arms: 1
Drug: Ibuprofen — Ibuprofen is given orally 600mg in the Post Anesthesia Care Unit, followed by an oral regime of 800mg twice a day
  Arms: 2
Drug: Acetaminophen — Acetaminophen is given 1g intravenously in the Operation room, followed by an oral regime of 1g fourth a day
  Arms: 3
Drug: Acetaminophen — Acetaminophen is given 1g intravenously in the operation room, followed by 1g orally fourth a day
  Arms: 3
Drug: Parecoxib/Valdecoxib — 40mg Parecoxib are given intravenously in the operation room, followed by 40mg of Valdecoxib orally twice a day
  Arms: 4
Other: Blood samples — Blood samples for aggregometry are taken before induction of anesthesia, 1h after first drug intake, 4hs and 24hs after first intake

SUMMARY:
Dipyrone is suggested to inhibit the platelet aggregation comparable to th effect of traditional analgetic substances like Ibuprofen. To verify this hypothesis the investigators conducted the study in comparing patients undergoing traumatologic, visceral or plastic surgical procedures. The investigators randomized them to four groups receiving common analgetic doses of either dipyrone, acetaminophen (paracetamol) or valdecoxib/parecoxib. The investigators took blood samples before initiation of the study drug, 1h, 4hs and 24hs after first intake. The investigators compared the aggregation via aggregometry of platelet rich plasma.

ELIGIBILITY:
Inclusion Criteria:

* Planned traumatologic, orthopedic, visceral or plastic surgical procedures

Exclusion Criteria:

* Prior intake of drugs with effect on the platelet aggregation
* Patients with diseases of the gastrointestinal systems
* Patients with cardiac or circulatory diseases
* Patients receiving corticoids
* Patients with cold or asthma
* ASA-classification > 3

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-02; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Percentage of aggregation in platelet rich plasma fter 24 hours of treatment with analgetic doses | 24 hours

SECONDARY OUTCOMES:
Percentage of aggregation of platelet rich plasma 1hour and 4 hours after initiation of study drug | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Schmauss, MD, Principal Investigator — research associate of the Ruhr University Bochum; Christoph Maier, Professor, Study Chair — Leader of the Department for Pain Medicine of the University Hospital Bergmannsheil Bochum
Locations (1):
- BG University Hospital Bergmannsheil GmbH, Bochum, Germany